CLINICAL TRIAL: NCT06694844
Title: Comparative Microbiome Analysis of Dental Biofilm on Two High-Density PTFE Membranes for Socket Preservation: A Molecular Evaluation of Streptococcus and Periodontopathogenic Species
Brief Title: Microbiome Analysis of Dental Biofilm on High-Density Polytetrafluoroethylene Membranes Used in Socket Preservation
Acronym: MADBioS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marija Čandrlić (Other)
Collaborators: University of Rijeka, Medical Faculty (Unknown); Clinical Hospital Center Rijeka (Other)
Responsible Party: Sponsor-Investigator, Marija Čandrlić, Faculty of Dental Medicine and Health, Josip Juraj Strossmayer University of Osijek
Organization: Josip Juraj Strossmayer University of Osijek (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2170/29-02/1-20-2
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Microbiology; Alveolar Ridge Preservation; Infections, Bacterial
Keywords: alveolar ridge preservation; non-resorbable membrane; guided bone regeneration; microbiology; dental biofilm; SEM; Next Generation Sequencing; RT-PCR
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M1 - permamem + bone grafting (Experimental): M1: In the group M1, the grafted site was covered with a d-PTFE membrane (Permamem®, botiss biomaterials GmbH, Zossen, Germany)
  Interventions: Procedure: Socket preservation with M1
- M2 - Cytoplast + bonegrafting (Active Comparator): • M2: In the group M2 the site was covered with an alternative d-PTFE membrane (Cytoplast™, Osteogenics Biomedical, Texas, USA)
  Interventions: Procedure: Socket preservation with M2

INTERVENTIONS:
Procedure: Socket preservation with M1 — Following extraction, socket will be filled with the combination of bovine xenograft and autograft and then covered with d-PTFE M1 membrane (peramem membrane).
  Arms: M1 - permamem + bone grafting
Procedure: Socket preservation with M2 — Following extraction, socket will be filled with the combination of bovine xenograft and autograft and then covered with d-PTFE M2 membrane (Cytoplast membrane).
  Arms: M2 - Cytoplast + bonegrafting

SUMMARY:
The goal of this clinical trial is to evaluate how different types of high-density polytetrafluoroethylene (d-PTFE) membranes impact dental biofilm accumulation and composition in patients undergoing socket preservation following tooth extraction. The main question it aims to answer are:

Does the type of d-PTFE membrane influence the diversity and composition of the dental biofilm in vivo? Therefore, the investigators will compare two types of d-PTFE membranes (Permamem® and Cytoplast™) to examine their respective effects on microbial colonization.

Participants will:

* Undergo tooth extraction followed by socket preservation with either the Permamem® or Cytoplast™ membrane, randomly assigned.
* Have biofilm samples collected from the membranes after 4 weeks for analysis through SEM, RT-PCR, and NGS methods.
* Return for follow-up visits, including a six-month check to evaluate healing progress and to continue with implant-prosthetics rehabilitation.

DETAILED DESCRIPTION:
This study was organized as a randomized controlled clinical trial, recruiting patients from a general population of oral surgery office. Participant are indicated for at least one tooth extraction and subsequent implant placement due to the failure of conventional therapies to preserve affected teeth. Before entering the study, all participants must provid informed consent after reviewing study details.

Out of 56 participants initially screened, 39 participants met the inclusion criteria and were randomly allocated to one of two study groups via a web-based randomization tool (https://www.randomizer.org/). In both groups, a socket grafting procedure will be performed immediately following tooth extraction, using a composite bone graft comprising 50% autogenous bone and 50% bovine xenograft (cerabone®, botiss biomaterials GmbH, Zossen, Germany), after the participants were randomly assigned to the following groups:

* M1: In the group M1, the grafted site was covered with a d-PTFE membrane (Permamem®, botiss biomaterials GmbH, Zossen, Germany), and
* M2: In the group M2 the grafted site was covered with an alternative d-PTFE membrane (Cytoplast™, Osteogenics Biomedical, Texas, USA).

No non-intervention control group was included in this study, as previous research studies have demonstrated that the absence of socket preservation leads to significantly greater volume loss compared to when preservation techniques are applied.

After tooth extraction and curettage, the integrity of the buccal bone wall will be assessed. Then, the base and central portion of the socket will be filled with autologous bone, while the remaining upper portion (up to the level of the buccal wall) will be filled with a 50:50 mixture of bovine bone biomaterial and autologous bone. A d-PTFE membrane will be positioned beneath the buccal and lingual soft tissue flaps, covering 3-5 mm of the upper bone wall. The central portion of the membrane will remain exposed, with no attempt to achive primary wound closure.

This approach allows for tailored membrane coverage based on the degree of buccal wall preservation, optimizing support for bone regeneration. Prior to surgery, all participants received mechanical plaque and calculus removal and were instructed in oral hygiene practices. An oral antibiotic Klavocin bid 1000 mg, Pliva, Zagreb, Croatia, or Clindamycin MIP 600 mg, Chem. Pharm. Fabrik GmbH, Ingbert, Germany, for penicillin-allergic patients, will be administered one hour before surgery. Additionally, patients rinsed with a 0.2% chlorhexidine digluconate solution (Parodontax 0.2%, Brentford, London, UK) preoperatively.

2.4. Surgical protocol and membrane extraction Following the preoperative assessment, local anesthesia 4% articaine hydrochloride with adrenaline at a concentration of 1:200,000 (Ubistesin Forte, 3M, Neuss, Germany) was administered to two regions: the area indicated for tooth extraction and the retromolar region in the same jaw quadrant, selected for autogenous bone harvesting. After atraumatic extraction of the tooth, the socket was thoroughly debrided, and the integrity of the bone walls was assessed with a periodontal probe (15 UNC Color-Coded, Hu-Friedy, Chicago, USA). Following an intrasulcular incision around the buccal surface of the adjacent teeth, a full-thickness mucoperiosteal flap was elevated using a surgical curette (Lucas 2.5 mm, Helmut Zepf, Seitingen-Oberflacht, Germany). Following a thorough assessment of the buccal bone walls and the required quantity of autograft, a full-thickness flap was elevated at the donor site, and autogenous bone was harvested using the Safescraper® Twist bone scraper (Geistlich Bone Harvesting Instruments, Basel, Switzerland). The donor site was subsequently closed with primary intention using standard suturing techniques.

The grafting was done with the mixture of bovine xenograft (cerabone®, Botiss Biomaterials GmbH, Zossen, Germany) and autograft. Based on group assignment, a d-PTFE membrane was used to cover the extraction socket - either permamem® (Botiss Biomaterials GmbH, Zossen, Germany) for the M1 group or Cytoplast™ (Osteogenics Biomedical, Texas, USA) for the M2 group. The flap was repositioned and secured with resorbable monofilament 6.0 sutures (SMI, St. Vith, Belgium, Surgicryl Rapid 6.0), leaving the central part of the membrane intentionally exposed.

Four weeks post-extraction, the d-PTFE membrane was removed in both groups, leaving the pseudoperiosteum covering the crestal part of the extraction socket exposed to support healing. The membrane was then prepared for further laboratory analysis, and healing was allowed to progress for six months, after which implant placement was performed in the prepared site.

To evaluate bacterial adherence on the d-PTFE membranes, samples were pre-pared for SEM analysis immediately after membrane removal following 4 weeks of healing. Following incubation in bacterial suspensions for 4 hours, the membranes were rinsed in sterile phosphate-buffered saline (PBS) and then air-dried in a high-flow sterile chamber. Membranes were then fixed at 4° C with a solution containing 4 % glutar-aldehyde and 0.5 % paraformaldehyde (Sigma-Aldrich, Burlington, Vermont, USA) in 0.1 M PBS (pH 7.2) (Sigma-Aldrich, Burlington, Vermont, USA). After fixation, samples underwent a graded dehydration process by immersion in increasing ethanol concen-trations (50%, 70%, 80%, 90%, and 100%) to prepare for imaging. Each membrane was then mounted onto a sample holder using conductive carbon tape. To enhance surface conductivity and prevent electron charging under the high-vacuum conditions of the electron beam, a thin 15 nm layer of gold-palladium was applied using the precision etching and coating system (PECS II, Gatan Inc., Pleasanton, California, USA). Finally, SEM imaging was conducted with a Jeol JSM-7800F field emission scanning electron microscope (JEOL Ltd., Tokyo, Japan), using an accelerating voltage of 7 kV and a working distance of 10 mm. This approach allowed for high-resolution visualization of biofilm morphology and bacterial distribution on the membrane surfaces.

Extraction of DNA nucleic acids DNA was isolated from collected membrane sonicate samples using the Nucleospin Tissue Kit (Macherey Nagel, Duren, Germany) following a modified bacterial protocol. Sonicated samples in 1.5 ml Eppendorf tubes were centrifuged at 15,000 rpm for 15 minutes, after which the supernatant was removed, leaving approximately 50 μl of sediment. This sediment was resuspended in 250 μl of a prepared G+ lysis buffer, as specified by the manufacturer's modified bacterial protocol, and vortexed thoroughly. Next, 40 μl of freshly prepared lysozyme solution was added, and the sample was incubated at 37°C for 1 hour. Following this, 30 μl of proteinase K was added, and the sample was incubated at 56°C for 2 hours. After incubation, 400 μl of B3 buffer was added, the sample was vortexed, and then incubated again at 70°C for 15 minutes. DNA was precipitated by adding 400 μl of chilled 98% ethanol. The manufacturer's protocol was resumed for subsequent steps, with the final elution volume reduced to 50 μl of BE. The concentration and purity of the extracted genomic DNA were assessed using a Qubit fluorometer.

Quantitative Real-Time PCR (qPCR) Analysis Quantification of bacteria in the membrane sonicate samples was performed using RT-PCR on an Applied Biosystems 7500 Fast Real-Time PCR System (Applied Biosystems, Foster City, California, USA), with specific TaqMan assays (Applied Biosystems, Foster City, California, USA) targeting key bacterial species. These assays included bacteria of cariogenic significance, such as the gram-positive facultative anaerobes Streptococcus mutans and Streptococcus sobrinus, known for their high-risk contribution to caries development, and Streptococcus salivarius, which acts as an antagonist to these species. Additionally, the gram-negative anaerobes Veillonella parvula and Aggregatibacter actinomycetemcomitans were analyzed to explore biofilm interactions and associations with gingival and periodontal infection progression. A specific TaqMan assay for the 16s rRNA gene was used to represent the total bacterial load in dental plaque. TaqMan assay primers and probes were designed to specifically target the genes for each bacteria. For total bacterial quantification, the conserved region of the 16s rRNA gene was selected as the reference.

The RT-PCR reaction mixture (20 µL) consisted of 10 µL of TaqMan Master Mix, 1 µL of individual Custom TaqMan assays for each selected bacterium, 4 µL of water, and 5 µL of DNA sample diluted to 0.5 ng/µL. Each TaqMan assay contained specific custom-designed primers for amplifying the gtfB, gtfT, tnpA, lktA, and rpoB genes, as well as the 16s rRNA gene as a reference control. Additionally, each assay included a custom-designed TaqMan fluorescently labeled probe with AM (fluorescein amidite) dye and a Q (quencher). The PCR conditions on the 7500 Fast Real-Time PCR System were as follows: an initial incubation at 95°C for 10 minutes for Taq DNA polymerase activation, followed by 50 cycles of 95°C for 15 seconds (DNA denaturation) and 60°C for 1 minute (primer binding and extension). The reactions were carried out in 96-well plates with triplicates for each bacterium, alongside non-template controls for all genes.

Detection and quantification of the amplified genes for each bacterial species and the total 16s rRNA were based on changes in the fluorescence signal of the TaqMan probes. Fluorescence was emitted upon hybridization and hydrolysis of the probe at the target nucleic acid site, so an increase in fluorescence intensity indicated the level of gene amplification. Results were measured using a threshold cycle (Ct) value, which represents the fluorescence level needed for detection and is consistently set within the exponential amplification phase. As sufficient DNA of the target gene is amplified, the fluorescent signal is detected, with the Ct value indicating the cycle in which detection occurred. A higher Ct value corresponds to a lower initial concentration of the target gene in the sample, while a lower Ct value indicates a higher initial concentration.

Relative quantification of each bacterial population was calculated using ΔCt, representing the difference between the Ct value for the target bacterial group and the Ct value for the total bacterial load (16s rRNA equivalent).

NGS For the purpose of amplicon sequencing of variable regions 3 and 4 of the 16S rRNA gene, DNA was isolated from the samples of 20 M1 and 16 M2 membranes and sent to the Molecular Research Laboratory (MRDNA) in Texas, USA. Amplicon sequencing used a set of primers 341F (5'-CCTAYGGGRBGCASCAG-3') and 806R (5'-GGACTACNNGGGTATCTAAT-3'). Sequencing data was downloaded from "Illumina's BaseSpace Sequence Hub" in the form of paired-end, demultiplexed fastq files. Data processing was performed using the software package Quantitative Insights Into Microbial Ecology 2 (QIIME2). Processing included filtering and denoising using the DADA2 program, concatenation of sequences (since pair-end sequencing was used), as well as the control for the presence of possible chimeras. For the taxonomic determination of microorganisms, the Naive Bayes classifier tool in QIIME2 was applied, adapted to work with the SILVA database, version 138. The sequences were grouped according to the criterion of 99% similarity.

The diversity and richness of all samples were estimated by alpha diversity (Shannon index) and beta diversity (Bray-Curtis dissimilarity) using the seaborn, matplotlib, pandas, and matplotlib libraries by Python programming language, version 3.12, within the Pycharm environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for tooth extraction due to:
* Deep caries lesions with chronic periapical periodontitis
* Fractures of the tooth crown and/or root
* Other conditions preventing conventional therapy
* Age between 18 and 60 years
* Physically and mentally healthy
* Patients who understand the study protocol and provide informed consent

Exclusion Criteria:

* Patients with any absolute contraindications for implant-prosthetic therapy (e.g., uncontrolled systemic diseases)
* Systemic conditions including:
* Uncontrolled diabetes
* Osteoporosis or osteopenia
* Vitamin D deficiency
* Patients on bisphosphonate or long-term glucocorticoid therapy
* Hypothyroidism
* Uncontrolled cardiovascular diseases (e.g., hypertension, coronary artery disease, congestive heart failure)
* Pregnant and lactating women

Local factors:

* Tobacco users (more than 10 cigarettes per day)
* Poor oral hygiene
* Patients with untreated periodontal disease
* History of radiation in the head and neck area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Scanning electron microscopy analaysis (SEM) | Up to 6 months
  Description: High-resolution imaging to visualize biofilm morphology and bacterial distribution on the membrane surfaces.
  Unit of Measure: Qualitative (e.g., bacterial morphology, density). Time Frame: Up to 6 months. This provides an observational outcome focused on the visual and qualitative analysis of biofilm structure.
RT-PCR | Up to 8 months
  Description: Quantitative analysis of specific bacterial species' presence and relative abundance associated with dental biofilm on d-PTFE membranes.
  Unit of Measure: Relative abundance (%) of targeted bacterial species. Time Frame: Up to 8 months. This measure captures the presence and amount of particular bacteria in biofilm samples.
Next Generation Sequencing (NGS) | Up to 10 months
  Description: Assessment of microbial diversity, richness, and specific bacterial composition on two types of d-PTFE membranes after a four-week healing period.
  Unit of Measure: Diversity indices (e.g., Shannon Index, species richness). Time Frame: Up to 10 months. This measure assesses the overall microbial community composition and diversity on each type of membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Cvijanovic Peloza, Full Professor, PhD, Study Chair — University of Rijeka, Faculty of Medicine
Locations (1):
- University of Rijeka, Faculty of Medicine Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon reasonable request after study results are published, solely for academic purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Around first quartal od 2025 to the end of 2028.
Access Criteria: Only academic stuff

REFERENCES:
- [Background] Begic G, Badovinac IJ, Karleusa L, Kralik K, Cvijanovic Peloza O, Kuis D, Gobin I. Streptococcus salivarius as an Important Factor in Dental Biofilm Homeostasis: Influence on Streptococcus mutans and Aggregatibacter actinomycetemcomitans in Mixed Biofilm. Int J Mol Sci. 2023 Apr 14;24(8):7249. doi: 10.3390/ijms24087249. PMID 37108414